CLINICAL TRIAL: NCT03966885
Title: Zambia Common Elements Treatment Approach Pilot Study
Acronym: ZCAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 precluded the study team from being able to complete all follow-up assessments.The study was halted on March 17, 2020 and did not resume.
Sponsor: Columbia University (Other)
Collaborators: Centre for Infectious Disease Research in Zambia (Other); University of Alabama at Birmingham (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jeremy C. Kane, Assistant Professor of Epidemiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAS7472; R34AA027200 (NIH)
Record Dates: First submitted 2019-05-23; First posted 2019-05-29 (Actual); Results first posted 2022-09-13 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Alcohol Use Disorder; Depression; Post-traumatic Stress Disorder; HIV/AIDS; Substance Use Disorders
MeSH Terms: conditions — Alcoholism; Depression; Stress Disorders, Post-Traumatic; Acquired Immunodeficiency Syndrome; Substance-Related Disorders | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Primary outcomes are evaluated via Audio Computer Assisted Self-Interviewing (ACASI)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Intervention (BI) (Experimental): 30 minute alcohol brief intervention delivered by lay provider during HIV clinic visit.
  Interventions: Behavioral: Brief Intervention
- Brief Intervention + CETA (Experimental): 30 minute alcohol brief intervention delivered by lay provider during clinic visit followed by 6-12 weekly sessions of CETA.
  Interventions: Behavioral: Brief Intervention; Behavioral: Common Elements Treatment Approach (CETA)

INTERVENTIONS:
Behavioral: Brief Intervention — The BI used in the trial combines motivational interviewing skills with cognitive behavioral therapy elements in order to assist clients with self identified substance misuse to begin to consider changing their rates of drinking and drug use. The intervention lasts 30 to 40 minutes and consists of 5 components including: 1) screening 2) identification and information on the impacts of substance misuse 3) talking about change and goal setting 4) understanding the primary reason for drinking 5) skill building with practice and 6) referral for services.
Behavioral: Common Elements Treatment Approach (CETA) — The Common Elements Treatment Approach, or CETA, is a transdiagnostic psychotherapy based on cognitive behavioral elements for mood, anxiety and trauma related problems, and for alcohol and substance misuse. CETA is based on the fact that most evidence-based mental health treatments (EBTs) consist of similar components. The objective of CETA is to provide a single training in a range of therapy components that are similar across EBTs and to then teach counselors how to design a specific course of treatment for each client based on the client's presenting problems.
  Arms: Brief Intervention + CETA

SUMMARY:
This is a randomized controlled trial (RCT) evaluating the effectiveness of an alcohol brief intervention alone compared to the brief intervention plus an evidence-based psychotherapy (CETA) in reducing alcohol misuse and co-occurring mental health problems among persons with HIV in Zambia.

DETAILED DESCRIPTION:
Alcohol misuse is a major unaddressed barrier to ending the HIV/AIDS epidemic. Hazardous drinking increases HIV transmission, delays antiretroviral therapy (ART) uptake, reduces adherence and retention, and increases mortality. Comorbid mental health or substance misuse, similar to alcohol use alone, can also significantly undermine HIV treatment. The vast majority of people living with HIV globally live in low- and middle-income countries (LMIC). Similar to most HIV care settings in LMIC, in Zambia, the location of the current study, there are no readily available evidence-based treatments for alcohol misuse or mental health problems.

This study will enroll persons living with HIV (PLWH) who have alcohol misuse in Zambia. Participants will be recruited and screened during regular HIV care visits. Participants will be recruited by their regular care providers (i.e., peer educators, counselors, nurses, physicians) and referred to study staff if they are interested. The investigators anticipate enrolling up to 320 participants, all of whom have hazardous alcohol use. N=160 participants will be high-risk drinkers due to having either a moderate-to-severe alcohol use disorder or mental health comorbidities, or both. These participants will be randomized into the RCT. Participants who have hazardous alcohol use (but not a moderate-to-severe AUD) without mental health comorbidities (a lower risk group of participants) will not be enrolled into the RCT but will be tracked as part of a parallel cohort study. The minimum age of research subjects will be 18. Eligibility will be assessed via audio computer assisted self-interviewing (ACASI).

Participants in the 'cohort study' (i.e., lower risk participants) will receive a brief alcohol intervention. Participants in the RCT (i.e., higher risk participants) will be randomly assigned on a 1:1 basis (stratified by gender) to receive the brief intervention alone or the brief intervention plus CETA.

All participants will be evaluated for outcomes at baseline and at a six month follow-up visit. For RCT participants, the investigators will compare the effectiveness of the brief intervention alone to the brief intervention plus CETA in reducing alcohol misuse and mental health problems. For cohort participants, the investigators will collect preliminary data on whether alcohol misuse reduced at the six month follow-up but there will be no comparison/control group.

The findings from this pilot study will be used to inform future programming and research in Zambia and other LMIC to implement screening, brief intervention, and referral to treatment (SBIRT) programs for alcohol use in HIV care.

ELIGIBILITY:
Inclusion Criteria:

* Initial inclusion criteria for overall enrollment (into either the Cohort or RCT study) will be:

  * HIV positive
  * Receiving HIV treatment services at one of the two study clinics
  * Current hazardous alcohol use, defined as an AUDIT score of ≥8 for men and ≥ 4 for women
  * Provides informed consent

Secondary inclusion for enrollment into the RCT will be:

* AUDIT scores that indicate a moderate-to-severe AUD (≥12 for women; ≥16 among men)
* AND/OR: meeting validated symptom criteria for depression (≥16 on Center for Epidemiological Studies-Depression (CES-D), trauma/anxiety (≥2.5 on HTQ), and/or substance use (≥27 for any non-tobacco/alcohol substance on ASSIST)

Exclusion Criteria:

* HIV negative
* Not receiving care at one of the study clinics
* Currently psychotic or actively suicidal
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy C. Kane, PhD, MPH, Principal Investigator — Columbia University
Locations (1):
- Centre for infectious Disease Research in Zambia, Lusaka, Zambia

REFERENCES:
- [Background] Kane JC, Sharma A, Murray LK, Chander G, Kanguya T, Lasater ME, Skavenski S, Paul R, Mayeya J, Kmett Danielson C, Chipungu J, Chitambi C, Vinikoor MJ. Common Elements Treatment Approach (CETA) for unhealthy alcohol use among persons with HIV in Zambia: Study protocol of the ZCAP randomized controlled trial. Addict Behav Rep. 2020 Apr 29;12:100278. doi: 10.1016/j.abrep.2020.100278. eCollection 2020 Dec. PMID 32637558
- [Result] Kane JC, Sharma A, Murray LK, Chander G, Kanguya T, Skavenski S, Chitambi C, Lasater ME, Paul R, Cropsey K, Inoue S, Bosomprah S, Danielson CK, Chipungu J, Simenda F, Vinikoor MJ. Efficacy of the Common Elements Treatment Approach (CETA) for Unhealthy Alcohol Use Among Adults with HIV in Zambia: Results from a Pilot Randomized Controlled Trial. AIDS Behav. 2022 Feb;26(2):523-536. doi: 10.1007/s10461-021-03408-4. Epub 2021 Jul 30. PMID 34328570

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brief Intervention (BI) | Brief Intervention + CETA
Started | 78 | 82
Completed | 56 | 62
Not Completed | 22 | 20
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 2
Not completed — Not post-assessed. Study ended early due to COVID-19 | 20 | 16
Not completed — Moved from study area. | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brief Intervention (BI) | Brief Intervention + CETA | Total
Number analyzed (Participants) | 78 | 82 | 160
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.8 (9) | 38.6 (9.4) | 40.2 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 36 | 70
  Male | 44 | 46 | 90
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 78 | 82 | 160
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Zambia | 78 | 82 | 160

OUTCOME MEASURES:

1. Primary Outcome: Change in Alcohol Use Disorders Identification Test (AUDIT) Scale Score From Baseline to 6-month Post-baseline.
Description: AUDIT is a 10-item measure of hazardous alcohol use with possible range of 0-40 (total scale score). Higher scores are associated with more hazardous use.
Time Frame: Baseline and 6 months post-baseline
Population: Analysis conducted only among participants with complete data at 6-month follow-up, which include 56 completers out of 78 participants in BI group and 62 completers out of 82 participants in BI + CETA group.
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Groups:
- Brief Intervention (BI): 30 minute alcohol brief intervention delivered by lay provider during HIV clinic visit.
  Brief Intervention (BI): The BI used in the trial combines motivational interviewing skills with cognitive behavioral therapy elements in order to assist clients with self identified substance misuse to begin to consider changing their rates of drinking and drug use. The intervention lasts 30 to 40 minutes and consists of 5 components including: 1) screening 2) identification and information on the impacts of substance misuse 3) talking about change and goal setting 4) understanding the primary reason for drinking 5) skill building with practice and 6) referral for services.
Arm/Group | Brief Intervention (BI) | Brief Intervention + CETA
Number analyzed (Participants) | 56 | 62
Score on a scale | -10.5 [-12.8 to -8.3] | -13.7 [-15.8 to -11.6]

2. Secondary Outcome: Change in Center for Epidemiological Studies-Depression (CES-D) Scale Score From Baseline to 6-month Post-baseline.
Description: CES-D is a 20-item scale of depression with a possible range of 0-60 (total scale score). Higher scores are associated with greater depression symptom severity.
Time Frame: Baseline and 6 months post-baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Brief Intervention (BI) | Brief Intervention + CETA
Number analyzed (Participants) | 56 | 62
Score on a scale | -4.2 [-7.2 to -1.1] | -8.9 [-11.8 to -6.0]

3. Secondary Outcome: Change in Harvard Trauma Questionnaire (HTQ) Post-traumatic Stress Disorder (PTSD) Symptom Scale Score From Baseline to 6-month Post-baseline.
Description: The HTQ is a 39-item PTSD symptom scale with possible range of 1-4 (average scale score). Higher scores are associated with greater PTSD symptom severity.
Time Frame: Baseline and 6 months post-baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Brief Intervention (BI) | Brief Intervention + CETA
Number analyzed (Participants) | 56 | 62
Score on a scale | -0.3 [-0.5 to -0.1] | -0.5 [-0.7 to -0.4]

4. Secondary Outcome: Number of Participants With Any Recent Substance Use.
Description: Any recent substance use will be defined as any use of the following substance types in the past 3 months: inhalants, marijuana, cocaine, amphetamines, sedatives, hallucinogens, opioids.
Time Frame: 6 months post-baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Brief Intervention (BI) | Brief Intervention + CETA
Number analyzed (Participants) | 56 | 62
Participants | 14 | 16

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Brief Intervention (BI) | Brief Intervention + CETA
All-Cause Mortality (participants affected / at risk) | 1/78 | 0/82
Serious Adverse Events (participants affected / at risk) | 1/78 | 0/82
Other Adverse Events (participants affected / at risk) | 0/78 | 0/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brief Intervention (BI) (N=78) | Brief Intervention + CETA (N=82)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Participant passed and the documented cause of death was reported as anemia, but it was not related to the intervention or study participation.

LIMITATIONS AND CAVEATS:
Study was stopped early due to COVID-19. Only participants who had completed their 6-month follow-up visit by March 17th, 2020 were included in analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/85/NCT03966885/Prot_SAP_000.pdf